CLINICAL TRIAL: NCT07359378
Title: Progressive Resistance Exercises Versus Functional Training in Elderly With Risk of Fall.
Brief Title: Progressive Resistance Exercise Versus Functional Training in Elderly With Risk of Fall.
Acronym: PRE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Haleema Imran, Dr., University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ethical review Board (IREB025)
Record Dates: First submitted 2025-12-26; First posted 2026-01-22 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Elderly
Keywords: fall; progressive resistive; functional training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study will implement single-blinding, where outcome assessors will remain unaware of group assignments to reduce assessment bias. Participants and session supervisors will not be blinded due to the nature of the interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Progressive Resistance Training
  Interventions: Other: Progressive Resistance Training
- Group 2 (Experimental): Functional Training
  Interventions: Other: Functional Training

INTERVENTIONS:
Other: Progressive Resistance Training — Intervention Protocol 1. Warm-Up (5 minutes) Gentle aerobic activities (marching in place, arm swings). Dynamic stretching to prepare muscles for resistance exercises. 2. Main Phase (35 minutes) Progressive resistance exercises targeting major muscle groups, applying the progressive overload principle (increasing resistance or repetitions biweekly). Exercises will include:
  o Lower body: Squats, seated leg press. o Upper body: Bicep curls, tricep extensions using dumbbells or resistance bands. o Core strengthening: Bridges. Focus on controlled movements and proper form to minimize injury risk. 19 3. Cooldown (5 minutes) Static stretching for major muscle groups to improve flexibility and promote recovery. (Coleman et al., 2021)
  Arms: Group 1
Other: Functional Training — 1. Warm-Up (5 minutes) Light walking in place, arm swings, and shoulder rolls to prepare the body. Dynamic stretching focusing on key muscle groups. 2. Main Phase (35 minutes) Exercises designed to enhance functional movements for daily activities: Sit-to-Stand (Chair Squats) - Strengthens legs and mimics standing up from a chair. Step-Ups - Improves leg strength and balance for climbing stairs. Heel-to-Toe Walk - Enhances balance and gait stability. Wall Push-Ups - Strengthens upper body for pushing movements. Bicep Curls with Resistance Bands - Improves arm strength for carrying objects. Ankle Circles - Enhances ankle mobility and balance. Progressive difficulty will be applied by increasing repetitions, reducing support, or adding light resistance. 3. Cooldown (5 minutes) 20 21 Gentle static stretching for major muscle groups. Breathing exercises for relaxation. (Ritterfeld et al., 2010)
  Arms: Group 2

SUMMARY:
Study Design: Randomized Clinical Trial Objective: To find the effects of Progressive Resistance Exercises for balance and risk of falls in elderly population.

To find the effects of Functional Training for balance and risk of falls in elderly population.

To compare the effects of Progressive Resistance Exercises and Functional Training for balance and risk of falls in elderly population.

Inclusion Criteria:

Both Males and Female Patients Patients Age 65 years or above Participants with intact cognitive function or mild cognitive impairment who can follow instructions and provide informed consent Individuals medically cleared by their physician to engage in moderate-intensity physical activities, with no unstable medical conditions that could impede participation Participants willing to commit to an 8-week intervention program (3 sessions per week) and attend follow-ups as required.

Exclusion Criteria:

Elderly individuals who are non-ambulatory or unable to perform basic mobility tasks, such as standing or walking independently, even with assistive devices.

Uncontrolled medical conditions such as uncontrolled hypertension, unstable angina, or severe arrhythmias.

Participants with severe musculoskeletal conditions that significantly limit mobility or exercise participation (e.g., severe arthritis, recent fractures, or joint replacements within the last 6 months).

Presence of acute pain or injury that may worsen with physical activity. Individuals with progressive neurological conditions such as Parkinson's disease, stroke with severe residual deficits, or multiple sclerosis that impede safe participation in physical activities.

Group 1: Progressive Resistance Exercises Participants in the Progressive Resistance Training (PRT) group will engage in a structured exercise program designed to progressively increase muscle strength, balance, and overall physical function.

Group 2: Functional Training Participants in the Functional Training (FT) group will engage in exercises that mimic daily activities to improve balance, strength, mobility, and functional independence.

DETAILED DESCRIPTION:
Study Design: Randomized Clinical Trial Settings: Study will be conducted at Shadman Medical centre and Jinnah Hospital, Lahore.

Duration of Study: The study will take 09 months after the approval of synopsis.

Sample Size:

The calculated sample size using TUG as an outcome measure is 33 in each group after adding 20% dropout the sample size will be 33+6=39 in each group.

Z1-α/2 Level of significance=95% µ1 Mean change in Group 1= 13 µ2 Mean change in Group 2= 16.7 s1 Standard deviation in group 1= 6.6 s2 Standard deviation in group 2= 3.6 Z1-β power of the study= 80% n sample size in a group= 33 After adding 20% drop out 33+6= 39 in each group.

Sampling Technique:

This study will employ a non-probability purposive sampling technique, ensuring the intentional selection of participants who meet specific inclusion criteria relevant to the study's focus on elderly individuals at risk of falls. This targeted approach enhances the study's relevance and validity by prioritizing individuals most likely to benefit from the interventions. To further ensure methodological rigor, participants will be randomly assigned to groups using a computer-generated randomization method, minimizing selection bias and balancing confounding variables. This combination of purposive sampling and random assignment ensures a robust and unbiased evaluation of the interventions under investigation.

SAMPLE SELECTION CRITERIA

Inclusion Criteria:

Both Males and Female Patients patients Age 65 years or above Participants with intact cognitive function or mild cognitive impairment who can follow instructions and provide informed consent Individuals medically cleared by their physician to engage in moderate-intensity physical activities, with no unstable medical conditions that could impede participation Participants willing to commit to an 8-week intervention program (3 sessions Per week) and attend follow-ups as required.

Exclusion Criteria:

Elderly individuals who are non-ambulatory or unable to perform basic mobility tasks, such as standing or walking independently, even with assistive devices.

Uncontrolled medical conditions such as uncontrolled hypertension, unstable angina, or severe arrhythmias.

Participants with severe musculoskeletal conditions that significantly limit mobility or exercise participation (e.g., severe arthritis, recent fractures, or joint replacements within the last 6 months).

Presence of acute pain or injury that may worsen with physical activity. Individuals with progressive neurological conditions such as Parkinson's disease, stroke with severe residual deficits, or multiple sclerosis that impede safe participation in physical activities.

ETHICAL CONSIDERATIONS

The research will adhere to the ethical guidelines established by the Institute Research Ethics Board (IREB) of the University of Lahore, ensuring that the rights and well-being of participants are upheld.

Written informed consent will be obtained from all participants and documented appropriately.

All details and statistics will be kept secret. Participants will be clearly informed that the study procedures pose no risks or disadvantages to them.

They will also be assured of their right to withdraw from the study at any stage without any repercussions.

All collected data and information will be treated with strict confidentiality Research participants will be notified about any physical, social, psychological and any other harm or danger due to study.

The effects of intervention will be explained to the participants. Participants will be ensured about the removal of their identity in any publication. We will protect their personal information at any cost.

Participants will be free to contribute to the study without any compulsion and will be able to leave the study at any time, we will respect their decision without any presssure on them to change their minds.

DATA COLLECTION PROCEDURE

SCREENING Participants will undergo a thorough screening process to ensure they meet the inclusion criteria while excluding conditions that could interfere with the study's outcomes. Screening will include a comprehensive medical history review, fall history, and baseline measurements such as age, BMI, and current physical activity levels. Tools like the Timed Up and Go (TUG) test, Berg Balance Scale (BBS) and FRAT(Falls risk assessment Tool) will be used at baseline to evaluate functional mobility, balance and risk of falls, respectively. This dual assessment will help establish participants' current balance deficit and risk of falls profiles.

RANDOMIZATION Eligible participants will be randomly assigned to one of two intervention groups-Progressive Resistance Training (Group 1) or Functional Training (Group 2)-using a computer-generated randomization technique. This method minimizes allocation bias, ensuring equal chances of assignment to either group.

BLINDING The study will implement single-blinding, where outcome assessors will remain unaware of group assignments to reduce assessment bias. Participants and session supervisors will not be blinded due to the nature of the interventions.

DEPENDENT AND INDEPENDENT VARIABLES

Dependent Variables:

oFunctional mobility (assessed using the Timed Up and Go (TUG) test). oBalance Assessment (assessed using the Berg Balance Scale (BBS)) oFall Risk Assessment (assessed using the FRAT)

Independent Variables:

oType of intervention (Progressive Resistance Training versus Functional Training).

INTERVENTIONS:

Group 1: Progressive Resistance Training Participants in the Progressive Resistance Training (PRT) group will engage in a structured exercise program designed to progressively increase muscle strength, balance, and overall physical function.

Baseline General Physiotherapy

Before starting the PRT program, participants will undergo general physiotherapy sessions, including:

Joint mobility exercises to improve flexibility. Basic balance training to assess stability. Functional movement drills to enhance coordination. Intervention Protocol

1. Warm-Up (5 minutes) Gentle aerobic activities (marching in place, arm swings). Dynamic stretching to prepare muscles for resistance exercises.
2. Main Phase (35 minutes) Progressive resistance exercises targeting major muscle groups, applying the progressive overload principle (increasing resistance or repetitions biweekly).

   Exercises will include:

   oLower body: Squats, seated leg press. oUpper body: Bicep curls, tricep extensions using dumbbells or resistance bands.

   oCore strengthening: Bridges. Focus on controlled movements and proper form to minimize injury risk.
3. Cooldown (5 minutes) Static stretching for major muscle groups to improve flexibility and promote recovery.

Group 2: Functional Training

Participants in the Functional Training (FT) group will engage in exercises that mimic daily activities to improve balance, strength, mobility, and functional independence.

Baseline General Physiotherapy

Before beginning the functional training program, participants will receive general physiotherapy, including:

Joint mobility exercises to improve flexibility. Basic balance training to assess postural stability. Gait and coordination drills to enhance walking mechanics. Functional Training Protocol

1. Warm-Up (5 minutes) Light walking in place, arm swings, and shoulder rolls to prepare the body. Dynamic stretching focusing on key muscle groups.
2. Main Phase (35 minutes)

   Exercises designed to enhance functional movements for daily activities:

   Sit-to-Stand (Chair Squats) - Strengthens legs and mimics standing up from a chair.

   Step-Ups - Improves leg strength and balance for climbing stairs. Heel-to-Toe Walk - Enhances balance and gait stability. Wall Push-Ups - Strengthens upper body for pushing movements. Bicep Curls with Resistance Bands - Improves arm strength for carrying objects. Ankle Circles - Enhances ankle mobility and balance. Progressive difficulty will be applied by increasing repetitions, reducing support, or adding light resistance.
3. Cooldown (5 minutes) Gentle static stretching for major muscle groups. Breathing exercises for relaxation.

ASSESSMENT:

Both groups will undergo baseline and post-intervention assessments to measure outcomes.

1. Timed Up and Go (TUG) Test:

   The TUG test will assess functional mobility and fall risk by recording the time taken to stand from a chair, walk three meters, turn around, and return to the chair.

   A time of >12 seconds will indicate an increased fall risk, providing an objective measure of dynamic balance and mobility.
2. Berg Balance Scale (BBS):

   The BBS will evaluate static and dynamic balance through 14 functional tasks, such as standing, reaching, turning, and stepping.

   Each task is scored on a 5-point ordinal scale (0-4), with a total score of 56. A score of ≤45 will indicate an increased risk of falls, providing a comprehensive measure of postural stability and balance control.
3. Fall Risk Assessment Tool (FRAT):

The FRAT is a screening tool used to identify individuals at risk of falling based on various intrinsic and extrinsic factors.

It consists of key components, including fall history, medication review, sensory deficits, and environmental hazards.

A scoring system categorizes individuals into low, moderate, or high risk for falls, guiding targeted intervention strategies.

The FRAT provides a comprehensive risk assessment by incorporating medical, functional, and environmental factors, aiding in fall prevention planning.

ELIGIBILITY:
Inclusion Criteria:

* Both Males and Female Patients
* Patients Age 65 years or above
* Participants with intact cognitive function or mild cognitive impairment who can follow instructions and provide informed consent
* Individuals medically cleared by their physician to engage in moderate-intensity physical activities, with no unstable medical conditions that could impede participation
* Participants willing to commit to an 8-week intervention program (3 sessions per week) and attend follow-ups as required.

Exclusion Criteria:

* Elderly individuals who are non-ambulatory or unable to perform basic mobility tasks, such as standing or walking independently, even with assistive devices.
* Uncontrolled medical conditions such as uncontrolled hypertension, unstable angina, or severe arrhythmias.
* Participants with severe musculoskeletal conditions that significantly limit mobility or exercise participation (e.g., severe arthritis, recent fractures, or joint replacements within the last 6 months).
* Presence of acute pain or injury that may worsen with physical activity. Individuals with progressive neurological conditions such as Parkinson's disease, 15 stroke with severe residual deficits, or multiple sclerosis that impede safe participation in physical activities.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-03-03 (Estimated); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale (BBS) | from enrollment to the end of treatment at 8 weeks
  The BBS will evaluate static and dynamic balance through 14 functional tasks, such as standing, reaching, turning, and stepping. Each task is scored on a 5-point ordinal scale (0-4), with a total score of 56. A score of ≤45 will indicate an increased risk of falls, providing a comprehensive measure of postural stability and balance control.

SECONDARY OUTCOMES:
Timed Up and Go Test | from enrollment till the end of treatment at 8 weeks
  The TUG test will assess functional mobility and fall risk by recording the time taken to stand from a chair, walk three meters, turn around, and return to the chair. A time of >12 seconds will indicate an increased fall risk, providing an objective measure of dynamic balance and mobility
Falls Risk Assessment Tool FRAT | From enrollment the end of treatment at 8 weeks
  The FRAT is a screening tool used to identify individuals at risk of falling based on various intrinsic and extrinsic factors. It consists of key components, including fall history, medication review, sensory deficits, and environmental hazards. A scoring system categorizes individuals into low, moderate, or high risk for falls, guiding targeted intervention strategies. 22 The FRAT provides a comprehensive risk assessment by incorporating medical, functional, and environmental factors, aiding in fall prevention planning.